CLINICAL TRIAL: NCT04923880
Title: Pragmatic Implementation Trial of a CF Primary Palliative Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: MJHS Institute for Innovation in Palliative Care (Other); Emory University (Other); Stony Brook University (Other); Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Anna M. Georgiopoulos, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P004090
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis; Quality of Life
Keywords: Palliative Care; Symptom Management
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: We have created a framework for a nationally generalizable model to improve best practices in generalist-level palliative care in CF. This framework links the screening approach of the CF Foundation Models of Palliative Care Guidelines to new sets of provider-level clinical best practice guides and practice-level processes of care, supported by targeted education and quality management. This protocol describes an implementation trial of this model that will rigorously evaluate its feasibility, uptake, and preliminary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of Primary Palliative Care Intervention in CF Centers (Other): Implement a Primary Palliative Care intervention comprising screening-and-triage workflows, best practice treatment guides for high frequency problems, patient/family and provider education, and a quality improvement (QI) toolkit in 5 CF centers.
  Interventions: Other: Implementation of Primary Palliative Care Intervention in CF Centers

INTERVENTIONS:
Other: Implementation of Primary Palliative Care Intervention in CF Centers — Individuals with CF ages 12 years and above will complete an annual palliative care needs assessment with the CF care team using the IPOS (Integrated Palliative Care Outcome Scale).
  Individuals with CF under 12 years of age will complete an annual palliative care needs assessment with the CF care team using IPOS as a conversation guide.
  Caregivers of Individuals with CF of all ages will be offered the BASC (Brief Assessment Scale for Caregivers).
  In addition to annual needs assessment, palliative care needs assessment will take place when triggered by changes in disease status, such as hospitalization, new diagnosis of CF related Diabetes or referral to transplant.

SUMMARY:
Five Cystic Fibrosis (CF) centers, key stakeholders, and a palliative care institute have collaborated to create a novel primary palliative care intervention for patients with CF, "Improving Life with CF: A Primary Palliative Care Partnership," and established the infrastructure and support necessary for a follow-on implementation study. This intervention provides a framework for a nationally generalizable model to improve best practices in generalist-level palliative care in CF.

Objectives:

Aim 1: Implement a primary palliative care intervention comprising screening-and-triage workflows, best practice treatment guides for high frequency problems, patient/family and provider education, and a quality improvement (QI) toolkit.

Aim 2: Evaluate feasibility, uptake, and preliminary outcomes during a multisite pragmatic, implementation trial of the intervention at 5 diverse Cystic Fibrosis (CF) Centers.

Subaim 2.1: Evaluate feasibility and uptake as measured by rates of screening and treatment delivery.

Hypothesis 1: Related to feasibility and uptake of the intervention:

1. > 80% of individuals with CF of all ages will receive an annual palliative care screening.
2. > 25% of individuals with CF will receive a palliative care screening prompted by hospitalization, new diagnosis of CF-Related Diabetes, need for transplantation, or another disease- or treatment-specific trigger.

Hypothesis 2: Related to provider education:

a) > 80% will access >1 training(s) (on-demand webinars or in-service by trained site educators).

Subaim 2.2: Evaluate data on preliminary outcomes for individuals with CF by comparing ratings on patient- and caregiver-reported outcome measures (e.g., Integrated Palliative Care Outcome Scale, Cystic Fibrosis Questionnaire-Revised, Memorial Symptom Assessment Scale-Cystic Fibrosis, and Brief Assessment Scale for Caregivers) during the trial to baseline ratings and exploring covariates of change (age, race/ethnicity, gender, disease severity, CFTR modifier treatment, psychological distress, and varied indicators reflecting intervention implementation).

DETAILED DESCRIPTION:
Introduction:

Palliative care is an interdisciplinary model of care intended to mitigate the suffering and illness burden experienced by patients with serious illnesses, and their families, from the time of diagnosis forward. The illness burden experienced by patients with CF and their caregivers is characterized by problems in many domains (e.g., physical symptoms, emotional distress, caregiver burden, and need for goal-setting). Interventions to address the goals of palliative care must be undertaken throughout the course of the illness by CF professionals-an approach known as generalist-level or primary palliative care. At present, there are no standardized, generalizable models of primary palliative care for CF.

New CF Foundation guidelines recommend that CF Centers screen all adults and children from the time of diagnosis, along with caregivers of individuals with CF of all ages, for unmet palliative care needs annually and after "triggers" such as hospitalization or other major events (Kavalieratos D et al. J Palliat Med. 2020 Sep 16. Epub ahead of print). The goal is to identify high frequency problems, such as symptom distress and the need for advance care planning (ACP).

The proposed intervention will involve a multi-site implementation trial of a new care model that applies the CF Foundation Palliative Care Guidelines (Kavalieratos D et al., 2020) at five CF Centers across the country. We will collect longitudinal data from patients and family caregivers on palliative care outcomes and also evaluate uptake of the care model.

Research conduct:

At baseline, each of the 5 participating CF Centers will recruit all eligible adolescent and adult CF patients plus one identified caregiver per patient of any age. Participants will have the opportunity to have their questions answered by a member of the site's study staff and will have at least 24 hours to decide whether they wish to participate. Those who agree to participate will be assigned a study ID number and their status tracked in a secure enrollment log.

Outcome Assessment:

Prior to the start of the system-level palliative care intervention involving individuals with CF and their primary caregivers at each site, patients and caregivers consenting to participate in the outcome assessment will complete a baseline questionnaire packet. This packet will include validated questionnaires that will be repeated during the outcome assessment. Participants will be reimbursed $20 for the baseline assessment, which is expected to take < 30 minutes to complete.

The baseline assessment will include sociodemographic items that assess age, gender, racial/ethnic status, primary language, marital status, educational level, employment status, annual household income, and insurance status, and will be completed by patients and caregivers to profile the cohort.

During the last 3 months of trial implementation, patients and caregivers who consented to participate in the baseline assessment will be asked to complete a second questionnaire packet (identical to the first). This will occur approximately 2 years following baseline, in study months 25-27. Participants will be reimbursed $20 for the outcome assessment, which is expected to take < 30 minutes to complete.

After the baseline research assessment, all study sites will seek to implement new CF Foundation guidelines recommending annual and triggered palliative care needs assessments for individuals with CF and their primary caregivers (Kavalieratos D et al., 2020). As each of the CF Centers in the study adopt this new system-wide care model, the proposed study will conduct an intervention trial to support practice change, involving: 1) practice-level screening-and-triage workflows, 2) best practice treatment guides for management of high frequency problems; 3) provider education in generalist-level palliative care, supported by on-demand webinars and 4) train-the-trainer approach (education and manuals); and 5) a QI toolkit including resources for patient and family education, the monitoring of quality indicators for successful implementation of routine screening, and focused studies related to specific objectives of palliative care.

Statistical Plan:

Process measures collected in the trial will include data on uptake of the intervention, including rates of screening, triage, use of best practice guides, and provider use of education (on-demand webinars and on-site in-services and training) at each site. For process measures, the electronic medical record or other tracking systems at each site will be queried quarterly under a waiver of written authorization for medical record abstraction. This de-identified, aggregate information, such as percentage of center patients who receive an annual or clinically triggered palliative care screening (e.g., Subaim 2.1, hypotheses 1a and 1b), will be entered by the Research Coordinator into a REDCap® database for the project.

All data from the participating sites (process data on intervention uptake from the electronic medical record, and quantitative data from patients and caregivers from REDCap®) will be merged into a SPSS database by the Research Manager at the Data Coordinating Center, MJHS Institute.

The process measures will provide information related to the feasibility and uptake of the proposed intervention. The analysis will evaluate a) the proportion of patients and caregivers who completed annual screenings vs. patients and caregivers who are eligible; b) the proportion of screenings completed by patients and caregivers following specific triggers: hospitalization, new diagnosis of CF-Related Diabetes, and referral/declined referral for transplant evaluation; c) the proportion of patients and caregivers whose screening identified a need for further assessment for various symptoms or needs; and d) the proportion of patients who underwent a change in care plan based on the triage approach for different symptoms or needs. The analysis will evaluate each of these outcomes by patient age group (adults, adolescents, older children, and young children). Uptake also will be assessed by the number of Care Team members who access on-demand webinars or on-site in-service training.

At each site, the new model will be judged to be feasible or not, based on whether the Center achieves all of the following benchmarks: 1) the structural components can be implemented and sustained over time and 2) by the outcome assessment, >80% of patients due for an annual screening are screened, and >25% of patients who need a 'triggered' screening are screened. The overall feasibility of the model relative to national distribution will be affirmed if at least four of the practices demonstrate that the model is feasible at the site.

This evaluation of feasibility will be complemented by exploratory quantitative analyses. In the quantitative analyses, all study variables will be described, and distributions evaluated. Generalized logistic linear mixed effects models will evaluate changes in all uptake variables. Uptake variables (1=screened, 0=not screened) will serve as the outcome in separate models.

All study variables will be described and distributions evaluated. Linear mixed effects models will evaluate changes in the typical primary outcomes (CFQ-R physical and emotional functioning subscale scores) and secondary outcomes (IPOS total score, MSAS-CF total score, total scores for the BASC, PHQ, GAD, PSS, and other CFQ-R subscales (e.g., vitality, digestive, respiratory symptoms, and role subscale scores)) as preliminary data for a fully-scaled randomized clinical trial. Time will serve as the fixed effect. Individual intercepts, site, and time will serve as random effects. The best fitting covariance structure will be selected using Akaike's Information Criterion. Additional separate models will evaluate patient- (sociodemographics, disease severity-, and psychological distress-related variables), provider- (use of education sessions), and site-level predictors of uptake (size of practice). SPSS version 25 will be used for all analyses. All analyses will be two-tailed with alpha set at .05. With baseline data prior to the intervention, longitudinal data from the outcome assessment, and process data about uptake of the intervention by each site, we also will be able to explore relationships between the intervention "dose" trends (e.g., the frequency of screening and triage across patients and the type of clinical interventions recommended and utilized) and effects on patient symptoms, function, or HRQL.

Monitoring and Quality Assurance:

Monitoring of source data will occur at each study site and by the Data Coordinating Center (the MJHS Institute). Process data on uptake of the intervention at the CF Centers and individual self-report or parent proxy report questionnaires, will be checked by research staff using a Standard Operating Procedure (SOP) Manual specifying the standard practices, methods, and protocol. A member of the study staff will cross-check all data and review all self-report measures to ensure their completeness. Any errors in completion will be reviewed to determine if directions or procedures for the assessments need to be altered. In this case, permission from the IRB will be requested to change any procedures. In addition, study personnel will use IRB-approved eligibility checklists to ensure that all patients and caregivers who are approached for participation in study assessments are eligible.

Research Coordinators at each site will be in weekly contact with the Site PIs and Research Manager at the Data Coordinating Center (the MJHS Institute) to review any issues with the data (i.e., missing data) and ensure data integrity. Given the multi-center nature of the study, the study PIs (Anna Georgiopoulos, MD, and Lara Dhingra, PhD) will also meet regularly by telephone and videoconference with the Site PIs to review study conduct at all sites. Sites will be required to review their progress regularly and report unanticipated events, protocol deviations, and protocol violations at least monthly to the study PIs.

Dr. Lara Dhingra, Co-PI at the MJHS Institute, the Data Coordinating Center for this study, and her research team will oversee the conduct of monthly protocol compliance audits. These will focus on informed consent procedures, participant eligibility, baseline and outcome assessments, and quarterly review of process measures. Protocol compliance will consist of 100% verification of the protocol specific measures identified in the protocol being available and accurately noted for the participant being reviewed. All study questionnaires will be audited for completeness by Dr. Dhingra, who also will conduct quality checks of the database that will receive this information; these data verification audits will be conducted for 100% of cases.

Safety Monitoring:

The proposed study has been reviewed by the Cystic Fibrosis Foundation Data Safety Monitoring Board, with the determination that the program is minimal risk and that there is no need for a Data Monitoring Committee for this study. Study PIs will be responsible for safety monitoring. Site PIs or their designees will be available at all times to respond to any question of safety.

ELIGIBILITY:
The primary palliative care intervention will be clinically implemented at a practice level at all CF centers and offered to all patients and families. For the baseline and outcome research questionnaire based surveys, inclusion and exclusion criteria are as follows:

Inclusion Criteria:

Patients (age > 12 years) who are treated at the participating CF Centers will be eligible for participation in the study if the following inclusion/exclusion criteria are met:

1. Have a diagnosis of CF.
2. Receive treatment at one of the participating CF Care Centers in the study.
3. Age ≥ 12 years.
4. For patients age 12-17 years, willingness and ability to provide implied informed consent by a parent or legal guardian for the patient's participation in the study, with child's implied assent, AND willingness and ability to provide consent by the parent or legal guardian for the parent's or guardian's participation in the caregiver assessment, for proxy completion of selected study measures.
5. For patients age >18 years, willingness and ability to provide implied informed consent for participation in the study.
6. Willingness to complete questionnaires two times.
7. English or Spanish as the primary language.
8. In order to ensure generalizability of the intervention, participants will not be excluded from the study for any of the following reasons:

   1. Extent of CF disease severity or lung/liver transplant status.
   2. Current use of CFTR modulators or other medical, psychological, or complementary therapies.
   3. Concomitant participation in another clinical research study.
   4. Lack of a participating caregiver for patients age > 18 years.

Caregivers (age > 18 years) will be eligible for participation if the following inclusion/exclusion criteria are met:

1. Are an identified caregiver of a patient with CF of any age, who receives treatment at one of the participating CF Care Centers in the study.

   1. For patients age < 18 years, the caregiver will be a parent or legal guardian.
   2. For patients age ≥ 18 years, the caregiver will be chosen by the patient (e.g., parent, spouse, partner, other relative or friend).
2. Willingness and ability to provide implied informed consent.
3. Willingness to complete questionnaires two times.
4. English or Spanish as the primary language.
5. The CF patient(s) (age > 12) for whom the caregiver provides CF care may accept or decline participation.

Exclusion Criteria:

Any subjects who are deemed unable to participate will be excluded, including those with evidence of cognitive impairment severe enough to prevent implied informed consent or completing the survey instruments, or at the PI's discretion.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals with CF receiving annual palliative care screening | 2 years
  Evaluate uptake of annual palliative care needs assessment process across 5 CF centers

SECONDARY OUTCOMES:
Proportion of individuals with CF receiving triggered palliative care screening | 2 years
  Evaluate uptake of palliative care needs assessment triggered by hospitalization, new diagnosis of CF-Related Diabetes, referral for transplantation, or another disease- or treatment-specific trigger across 5 CF centers
Use of primary palliative care provider education materials | 2 years
  Proportion of CF healthcare providers who access 1 or more on-demand webinars or in-service trainings across 5 CF centers
Integrated Palliative Care Outcome Scale (IPOS) | 2 years
  multidimensional palliative care needs
Memorial Symptom Assessment Scale-Cystic Fibrosis (MSAS-CF) | 2 years
  symptom burden
Cystic Fibrosis Questionnaire-Revised (CFQ-R) | 2 years
  health-related quality of life
Patient Health Questionnaire-8 (PHQ-8) | 2 years
  depressive symptoms
Generalized Anxiety Disorder-7 item Scale (GAD-7) | 2 years
  anxiety symptoms
PROMIS® Parent Proxy Anxiety-Short Form (PASF) | 2 years
  anxiety symptoms
PROMIS® Parent Proxy Depression-Short Form (PDSF) | 2 years
  depression symptoms
PROMIS® Parent Proxy Pain Interference-Short Form 8a (PPISF) | 2 years
  pain interference
Perceived Stress Scale (PSS) | 2 years
  patient/caregiver stress
PROMIS® Global Health-Short Form (PGHSF) | 2 years
  caregiver quality of life
Brief Assessment Scale for Caregivers (BASC) | 2 years
  caregiver burden

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Georgiopoulos, MD, Principal Investigator — Massachusetts General Hospital (MGH); Lara Dhingra, PhD, Principal Investigator — MJHS Institute for Innovation in Palliative Care (MJHS Institute)
Locations (5):
- United States (5):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Northwell Health-Lenox Hill, New York, New York
  - Northwell Health, New York, New York
  - Stonybrook University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The dataset for this study, including the study protocol, statistical analysis plan, and individual de-identified participant data underlying the results reported in publication (text, tables, figures and appendices), will be made accessible four months from initial request to investigators who provide a methodologically sound proposal, as determined by the study's lead investigators. The dataset will be provided after its de-identification, in compliance with relevant regulatory and privacy laws, data safeguards, and requirements for patient consent and anonymization.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months after study publication.
Access Criteria: Investigators submitting a methodologically sound proposal, as determined by the study's lead investigators. Proposals should be directed to ldhingra@mjhs.org.

REFERENCES:
- [Background] Dhingra L, Walker P, Berdella M, Plachta A, Chen J, Fresenius A, Balzano J, Barrett M, Bookbinder M, Wilder K, Glajchen M, Langfelder-Schwind E, Portenoy RK. Addressing the burden of illness in adults with cystic fibrosis with screening and triage: An early intervention model of palliative care. J Cyst Fibros. 2020 Mar;19(2):262-270. doi: 10.1016/j.jcf.2019.08.009. Epub 2019 Aug 27. PMID 31471264
- [Background] Dellon EP, Goggin J, Chen E, Sabadosa K, Hempstead SE, Faro A, Homa K. Defining palliative care in cystic fibrosis: A Delphi study. J Cyst Fibros. 2018 May;17(3):416-421. doi: 10.1016/j.jcf.2017.10.011. Epub 2017 Oct 31. PMID 29097163
- [Background] Quill TE, Abernethy AP. Generalist plus specialist palliative care--creating a more sustainable model. N Engl J Med. 2013 Mar 28;368(13):1173-5. doi: 10.1056/NEJMp1215620. Epub 2013 Mar 6. No abstract available. PMID 23465068
- [Background] Kavalieratos D, Georgiopoulos AM, Dhingra L, Basile MJ, Rabinowitz E, Hempstead SE, Faro A, Dellon EP. Models of Palliative Care Delivery for Individuals with Cystic Fibrosis: Cystic Fibrosis Foundation Evidence-Informed Consensus Guidelines. J Palliat Med. 2021 Jan;24(1):18-30. doi: 10.1089/jpm.2020.0311. Epub 2020 Sep 16. PMID 32936045
- [Background] Georgiopoulos AM, Friedman D, Porter EA, Krasner A, Kakarala SP, Glaeser BK, Napoleon SC, Wozniak J. Screening for ADHD in adults with cystic fibrosis: Prevalence, health-related quality of life, and adherence. J Cyst Fibros. 2018 Mar;17(2):276-280. doi: 10.1016/j.jcf.2017.08.011. Epub 2017 Sep 1. PMID 28867260
- [Background] Quittner AL, Goldbeck L, Abbott J, Duff A, Lambrecht P, Sole A, Tibosch MM, Bergsten Brucefors A, Yuksel H, Catastini P, Blackwell L, Barker D. Prevalence of depression and anxiety in patients with cystic fibrosis and parent caregivers: results of The International Depression Epidemiological Study across nine countries. Thorax. 2014 Dec;69(12):1090-7. doi: 10.1136/thoraxjnl-2014-205983. Epub 2014 Sep 21. PMID 25246663
- [Background] Linnemann RW, O'Malley PJ, Friedman D, Georgiopoulos AM, Buxton D, Altstein LL, Sicilian L, Lapey A, Sawicki GS, Moskowitz SM. Development and evaluation of a palliative care curriculum for cystic fibrosis healthcare providers. J Cyst Fibros. 2016 Jan;15(1):90-5. doi: 10.1016/j.jcf.2015.03.005. Epub 2015 Mar 25. PMID 25817162
- [Background] Friedman D, Linnemann RW, Altstein LL, Islam S, Bach KT, Lamb C, Volpe J, Doolittle C, St John A, O'Malley PJ, Sawicki GS, Georgiopoulos AM, Yonker LM, Moskowitz SM. The CF-CARES primary palliative care model: A CF-specific structured assessment of symptoms, distress, and coping. J Cyst Fibros. 2018 Jan;17(1):71-77. doi: 10.1016/j.jcf.2017.02.011. Epub 2017 Mar 14. PMID 28302366
- [Background] Friedman D, Linnemann RW, Altstein LL, Georgiopoulos AM, Islam S, Bach KT, St John A, Fracchia MS, Neuringer I, Lapey A, Sicilian L, Moskowitz SM, Yonker LM. Effects of a primary palliative care intervention on quality of life and mental health in cystic fibrosis. Pediatr Pulmonol. 2019 Jul;54(7):984-992. doi: 10.1002/ppul.24311. Epub 2019 Mar 10. PMID 30854795
- [Background] Linnemann RW, Friedman D, Altstein LL, Islam S, Bach KT, Georgiopoulos AM, Moskowitz SM, Yonker LM. Advance Care Planning Experiences and Preferences among People with Cystic Fibrosis. J Palliat Med. 2019 Feb;22(2):138-144. doi: 10.1089/jpm.2018.0262. Epub 2018 Oct 18. PMID 30335569
- [Background] Balzano J, Fresenius A, Walker P, Berdella M, Portenoy RK, Bookbinder M, Glajchen M, Plachta A, Langfelder-Schwind E, Chen J, Dhingra L. Web-based symptom screening in cystic fibrosis patients: A feasibility study. J Cyst Fibros. 2016 Jan;15(1):102-8. doi: 10.1016/j.jcf.2015.11.001. Epub 2015 Nov 21. PMID 26610859
- [Background] Wojtaszczyk A, Glajchen M, Portenoy RK, Berdella M, Walker P, Barrett M, Chen J, Plachta A, Balzano J, Fresenius A, Wilder K, Langfelder-Schwind E, Dhingra L. Trajectories of caregiver burden in families of adult cystic fibrosis patients. Palliat Support Care. 2018 Dec;16(6):732-740. doi: 10.1017/S1478951517000918. Epub 2017 Oct 17. PMID 29037271
- [Background] Ahluwalia SC, Chen C, Raaen L, Motala A, Walling AM, Chamberlin M, O'Hanlon C, Larkin J, Lorenz K, Akinniranye O, Hempel S. A Systematic Review in Support of the National Consensus Project Clinical Practice Guidelines for Quality Palliative Care, Fourth Edition. J Pain Symptom Manage. 2018 Dec;56(6):831-870. doi: 10.1016/j.jpainsymman.2018.09.008. Epub 2018 Oct 31. PMID 30391049
- [Background] Basile M, Jojan L, Hobler MR, Dellon EP, Georgiopoulos AM, Goggin JL, Chen E, Goss CH, Hempstead SE, Faro A, Kavalieratos D. Assessing Practices, Beliefs, and Attitudes about Palliative Care among People with Cystic Fibrosis, Their Caregivers, and Clinicians: Results of a Content Analysis. J Palliat Med. 2021 Nov;24(11):1650-1656. doi: 10.1089/jpm.2020.0725. Epub 2021 Apr 20. PMID 33885355
- [Background] Collins ES, Witt J, Bausewein C, Daveson BA, Higginson IJ, Murtagh FE. A Systematic Review of the Use of the Palliative Care Outcome Scale and the Support Team Assessment Schedule in Palliative Care. J Pain Symptom Manage. 2015 Dec;50(6):842-53.e19. doi: 10.1016/j.jpainsymman.2015.07.015. Epub 2015 Aug 31. PMID 26335764
- [Background] Sawicki GS, Sellers DE, Robinson WM. Self-reported physical and psychological symptom burden in adults with cystic fibrosis. J Pain Symptom Manage. 2008 Apr;35(4):372-80. doi: 10.1016/j.jpainsymman.2007.06.005. Epub 2008 Jan 22. PMID 18215497
- [Background] Collins JJ, Devine TD, Dick GS, Johnson EA, Kilham HA, Pinkerton CR, Stevens MM, Thaler HT, Portenoy RK. The measurement of symptoms in young children with cancer: the validation of the Memorial Symptom Assessment Scale in children aged 7-12. J Pain Symptom Manage. 2002 Jan;23(1):10-6. doi: 10.1016/s0885-3924(01)00375-x. PMID 11779663
- [Background] Collins JJ, Byrnes ME, Dunkel IJ, Lapin J, Nadel T, Thaler HT, Polyak T, Rapkin B, Portenoy RK. The measurement of symptoms in children with cancer. J Pain Symptom Manage. 2000 May;19(5):363-77. doi: 10.1016/s0885-3924(00)00127-5. PMID 10869877
- [Background] Modi AC, Quittner AL. Validation of a disease-specific measure of health-related quality of life for children with cystic fibrosis. J Pediatr Psychol. 2003 Dec;28(8):535-45. doi: 10.1093/jpepsy/jsg044. PMID 14602844
- [Background] Quittner AL, Sawicki GS, McMullen A, Rasouliyan L, Pasta DJ, Yegin A, Konstan MW. Erratum to: Psychometric evaluation of the Cystic Fibrosis Questionnaire-Revised in a national, US sample. Qual Life Res. 2012 Sep;21(7):1279-90. doi: 10.1007/s11136-011-0091-5. Epub 2012 Jan 13. PMID 22240933
- [Background] Quittner AL, Schechter MS, Rasouliyan L, Haselkorn T, Pasta DJ, Wagener JS. Impact of socioeconomic status, race, and ethnicity on quality of life in patients with cystic fibrosis in the United States. Chest. 2010 Mar;137(3):642-50. doi: 10.1378/chest.09-0345. Epub 2009 Oct 9. PMID 19820076
- [Background] Quittner AL, Modi AC, Wainwright C, Otto K, Kirihara J, Montgomery AB. Determination of the minimal clinically important difference scores for the Cystic Fibrosis Questionnaire-Revised respiratory symptom scale in two populations of patients with cystic fibrosis and chronic Pseudomonas aeruginosa airway infection. Chest. 2009 Jun;135(6):1610-1618. doi: 10.1378/chest.08-1190. Epub 2009 May 15. PMID 19447923
- [Background] Alpern AN, Brumback LC, Ratjen F, Rosenfeld M, Davis SD, Quittner AL. Initial evaluation of the Parent Cystic Fibrosis Questionnaire--Revised (CFQ-R) in infants and young children. J Cyst Fibros. 2015 May;14(3):403-11. doi: 10.1016/j.jcf.2014.11.002. Epub 2014 Nov 28. PMID 25443473
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Pilkonis PA, Yu L, Colditz J, Dodds N, Johnston KL, Maihoefer C, Stover AM, Daley DC, McCarty D. Item banks for alcohol use from the Patient-Reported Outcomes Measurement Information System (PROMIS): use, consequences, and expectancies. Drug Alcohol Depend. 2013 Jun 1;130(1-3):167-77. doi: 10.1016/j.drugalcdep.2012.11.002. Epub 2012 Dec 1. PMID 23206377
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Golden-Kreutz DM, Browne MW, Frierson GM, Andersen BL. Assessing stress in cancer patients: a second-order factor analysis model for the Perceived Stress Scale. Assessment. 2004 Sep;11(3):216-23. doi: 10.1177/1073191104267398. PMID 15358877
- [Background] Irwin DE, Gross HE, Stucky BD, Thissen D, DeWitt EM, Lai JS, Amtmann D, Khastou L, Varni JW, DeWalt DA. Development of six PROMIS pediatrics proxy-report item banks. Health Qual Life Outcomes. 2012 Feb 22;10:22. doi: 10.1186/1477-7525-10-22. PMID 22357192
- [Background] Scott EL, Foxen-Craft E, Caird M, Philliben R, deSebour T, Currier E, Voepel-Lewis T. Parental Proxy PROMIS Pain Interference Scores are Only Modestly Concordant With Their Child's Scores: An Effect of Child Catastrophizing. Clin J Pain. 2020 Jan;36(1):1-7. doi: 10.1097/AJP.0000000000000772. PMID 31599745
- [Background] Glajchen M, Kornblith A, Homel P, Fraidin L, Mauskop A, Portenoy RK. Development of a brief assessment scale for caregivers of the medically ill. J Pain Symptom Manage. 2005 Mar;29(3):245-54. doi: 10.1016/j.jpainsymman.2004.06.017. PMID 15781175
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- See also: Science of Behavior change: Parent Related stress (NIH perceived scale) — https://scienceofbehaviorchange.org/measures/parent-rated-stress-nih-perceived-stress-scale/?id=0
- See also: Palliative care outcome scale — https://pos-pal.org/